CLINICAL TRIAL: NCT02890953
Title: Efficacy and Safety Evaluation of Pneumostem® Versus a Control Group for Treatment of IVH in Premature Infants (Phase 2a)
Brief Title: Efficacy and Safety of Pneumostem® for IVH in Premature Infants (Phase 2a)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Won Soon Park, Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2016-06-005
Record Dates: First submitted 2016-08-31; First posted 2016-09-07 (Estimated); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Cell Transplantation
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Placebo Comparator): Control group receives placebo medication (normal saline)
  Interventions: Drug: Normal saline
- MSC group (Experimental): MSC group receives mesenchymal stem cells transplantation (Pneumostem)
  Interventions: Drug: Pneumostem

INTERVENTIONS:
Drug: Pneumostem — direct intracerebroventricular injection of mesenchymal stem cells via ventricular tap
  Other Names: Umbilical cord blood derived mesenchymal stem cells
  Arms: MSC group
Drug: Normal saline — direct intracerebroventricular injection of normal saline via ventricular tap
  Arms: Control

SUMMARY:
The objective of this study is to evaluate the efficacy and safety of a single intraventricular administration of Pneumostem® for treatment of Intraventricular hemorrhage (IVH) in high-risk premature infants by comparing Pneumostem-treated group with a control group.

ELIGIBILITY:
Inclusion Criteria:

* IVH grade 3-4
* age : within postnatal day 28
* gestational age: 23-<34 weeks

Exclusion Criteria:

* Patient with severe congenital abnormalities
* Patient with antenatal brain hemorrhage
* Patient with asphyxia or Hypoxic ischemic encepalophathy
* Patient with chromosome anomalies (i.e. Edward syndrome, Patau syndrome, Down syndrome, etc) or severe congenital malformation (Hydrocephalus, Encephalocele, etc)
* Patient with a concurrent severe congenital infection (i.e. Herpes, Toxoplasmosis, Rubella, Syphilis, AIDS, etc)
* Patient withCRP > 30 mg/dL; Severe sepsis or shock
* Patient with a history of participating in other clinical studies
* Patient who is considered inappropriate to participate in the study by the investigator

Max Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Estimated)
Dates: Start 2017-03-28 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Shunt or death | 40 weeks of corrected age
  Shunt operation or death

SECONDARY OUTCOMES:
Death | at 2years
  Death
Developmental delay in gross motor function, 2y | at 2years
  Cerebral palsy, gross motor function classification system score ≥2
Developmental delay Bayley -3 | at 2years
  Bayley-3 scores <70
Developmental delay in KDST, 2y | at 2 years
  Korean Developmental Screening Test scores, below two standard deviations was classified as delayed
Language delay | at 2 years, at 5 years
  Korean Sequenced Language Scale for Infant score
Developmental delay in KDST, 5y | at 5 years
  Korean Developmental Screening Test scores, below two standard deviations was classified as delayed
Developmental delay in gross motor function | at 2years
  Cerebral palsy, gross motor function classification system score ≥2
Developmental delay in gross motor function, 5y | at 5years
  Cerebral palsy, gross motor function classification system score ≥2
epilepsy | at 2 years, at 5 years
  epilepsy required anti-seizure medication or treatment

CONTACTS AND LOCATIONS:
Overall Officials: So Yoon Ahn, MD. Ph.D, Study Director — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No